CLINICAL TRIAL: NCT05531929
Title: Study of the Role of Anxiety-related Antecedents on the Resumption of Work and Sport in a Series of Patients Operated on for Rotator Cuff Repair
Brief Title: Role of Anxio-depressive History on Return to Work and Sport After Rotator Cuff Surgery
Acronym: Reprise
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8614
Record Dates: First submitted 2022-09-02; First posted 2022-09-08 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Anxiety Depression Disorder
Keywords: Anxiety Depression Disorder; Rotator cuff repair

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Anxiety-depressive disorders are also very frequent, in the form of different pathologies that are often intertwined (prevalence of generalized anxiety disorders in 5% of the population, characterized depressive episodes in 5%, etc.).

And it is even more frequent in patients with a cuff tendinopathy (26% and 23% of depression and anxiety respectively). These 2 pathologies are therefore responsible for significant economic expenses.

It is in this context that the investigators' wish to carry out this study seems justified in order to better understand and therefore manage this problem, which is frequently encountered in daily practice and which would therefore allow better understanding and therefore better information for the patients concerned.

ELIGIBILITY:
Inclusion criteria:

* Major subject (≥ 18 years)
* Operated between January 2008 and September 2009 arthroscopically for a symptomatic supraspinatus tendon rupture, retracted in zone 1, resistant to medical treatment with a mobile shoulder, fatty degeneration of stage 2 or less with also a preserved subacromial space
* Subject not objecting to the reuse of their data for scientific research purposes.

Exclusion criteria:

- Subject having expressed his opposition to the reuse of his data for scientific research purposes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Major subject (≥ 18 years) operated between January 2008 and September 2009 arthroscopically for a symptomatic supraspinatus tendon rupture
Sampling Method: Non-Probability Sample
Enrollment: 212 (Actual)
Dates: Start 2022-05-22 (Actual); Primary Completion 2022-10-22 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
Measurement of the duration of complete sports cessation after rotator cuff repair surgery | 6 months after rotator cuff repair surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Chirurgie orthopédique de l'épaule et du coude - CHU de Strasbourg - France, Strasbourg, France